CLINICAL TRIAL: NCT04028583
Title: Tool for Inappropriate Prescription Evaluation: The TaIPE Study
Acronym: TaIPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Chantal Csajka, Principal Investigator, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TaIPE
Record Dates: First submitted 2019-07-17; First posted 2019-07-22 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Inappropriate Prescribing
Keywords: Inappropriate Prescribing; Potentially Inappropriate Medication List; Aged; Practice Guideline; Education, Medical
MeSH Terms: interventions — Potentially Inappropriate Medication List

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PIM-Check group (Experimental)
  Interventions: Other: PIM-Check
- STOPP/START group (Active Comparator)
  Interventions: Other: STOPP/START

INTERVENTIONS:
Other: PIM-Check — In the PIM-Check group, a medication review will be conducted using PIM-Check within 72 hours of patient's admittance to the unit. The physician will decide whether to accept these recommendations or not and implement prescribing changes if agreed.
  Arms: PIM-Check group
Other: STOPP/START — In the STOPP/START group, medication lists will be analyzed within 72 hours of patient's admittance and optimized according to STOPP/START criteria. The second physician will decide whether to accept these recommendations or not and implement prescribing changes if agreed.
  Arms: STOPP/START group

SUMMARY:
A mono-center, randomized controlled trial will be conducted at the University Hospital of Lausanne. Hospitalized patients will be randomly assigned from the emergency department to two sub-units composing the acute care for elders (ACE) unit. In one subunit, potentially inappropriate prescriptions will be detected and treatment optimized according PIM-Check. In the other, STOPP/START criteria will be independently applied.

ELIGIBILITY:
Inclusion Criteria:

* All patients meeting the admission criteria of the acute care for elders (ACE) unit will be eligible.

Exclusion Criteria:

* none

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 464 (Estimated)
Dates: Start 2018-02-26 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-08-04 (Estimated)

PRIMARY OUTCOMES:
Rate of Potentially Inappropriate Prescriptions (PIPs) reduction in the PIM-Check group compared to STOPP/START | 18 months

SECONDARY OUTCOMES:
Number and type of PIPs detected by each tool | 18 months
Rate of acceptability | 18 months
Number of treatment (mean and median) modification by clinicians | 18 months
Number of drugs at discharge | 18 months
Incidence rate of falls | 18 months
Activities of daily living (ADL) score | 18 months
  Activities of daily living are routine activities people do every day without assistance (6 basic activities) : eating, bathing, getting dressed, toileting, transferring, and continence. The score is the number of activities performed without assistance. Score ranges : from 0/6 (minimum) to 6/6 (maximum). Higher values represent a better outcome of activities of daily living.
Confusion Assessment Method (CAM) | 18 months
  Result ranges : [negative result (-) = no confusion] ; [positive result (+) = confusion].
Length of stay | 18 months
Number of unplanned readmission | up to 3 months after discharge
Association between the number and type of PIPs at discharge with rate of re-admission | up to 3 months after discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Farhat A, Al-Hajje A, Lang PO, Csajka C. Impact of Pharmaceutical Interventions with STOPP/START and PIM-Check in Older Hospitalized Patients: A Randomized Controlled Trial. Drugs Aging. 2022 Nov;39(11):899-910. doi: 10.1007/s40266-022-00974-7. Epub 2022 Sep 30. PMID 36175740